CLINICAL TRIAL: NCT03129919
Title: Arch Dimension and Inclination of the Upper and Lower Incisors Changes in Patients Treated With Interactive and Passive Self-ligation Brackets
Brief Title: Arch Dimension and Inclination of the Upper and Lower Incisors Changes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Principal Investigator, Claudia Vivian Forero Manrique, Self-ligating clinical professor, Fundación Universitaria CIEO
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2017-03-22; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Malocclusion, Angle Class I
MeSH Terms: conditions — Malocclusion, Angle Class I

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orthodontic patients treated with brackets Carriere SLX® (Experimental): Subjects requiring orthodontic treatment and will be treated with passive self-ligating braces Carriere SLX®
  Interventions: Device: Carriere SLX® (Passive self-ligating braces)
- Orthodontic patients treated with brackets Empower® (Active Comparator): Subjects requiring orthodontic treatment and will be treated with interactive self-ligating braces Empower®
  Interventions: Device: Empower® (Interactive self-ligating braces)

INTERVENTIONS:
Device: Carriere SLX® (Passive self-ligating braces) — Changes in the inclination of the incisors, expansion of the arches at the end of the alignment and leveling phase of the orthodontic treatment
  Arms: Orthodontic patients treated with brackets Carriere SLX®
Device: Empower® (Interactive self-ligating braces) — Changes in the inclination of the incisors, expansion of the arches at the end of the alignment and leveling phase of the orthodontic treatment
  Arms: Orthodontic patients treated with brackets Empower®

SUMMARY:
It is intended to evaluate changes in arch dimensions and incisor inclination as well as changes in the WALA Ridge in no extraction patients treated with interactive self-ligating brackets (Empower®) and passive (Carriere SLX®) at the end of the phase of alignment and leveling. For this, study models and profile radiographs taken before the start of treatment and at the end of the alignment and leveling phase will be evaluated. The parameters to be measured are: intercanine distance, arch depth, upper and lower incisor inclination, and WALA ridge analysis

ELIGIBILITY:
Inclusion Criteria:

* Complete permanent dentition, except third molars.
* Class I malocclusion, determined by Angle ANB 2 plus or minus 2
* Visible alveolar teeth and ridges in plaster models, the latter being compatible and checked against the morphology of the WALA Ridge clinically presented by the patient.
* Little index with minimum Irregularity 4-6 mm.
* Patients with x-rays of initial profile and at the end of alignment and leveling in good condition.

Exclusion Criteria:

* Models in poor condition that do not allow measurements.
* Patients who do not wish to participate in the study
* Patients with cleft lip and palate
* Patients with craniofacial anomalies
* Patients with previous orthodontic treatment

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
Incisomaxillary angle | At the end of the alignment and leveling phase, an average of 8 months
  Angle formed by the palatal plane and the upper incisor

SECONDARY OUTCOMES:
Transverse development of the upper and lower jaws | Each time wire is changed in the sequence suggested by the author, an average of 3 months
  Cuspal and basal intercanine distance
Inclination of the lower incisor | At the end of the alignment and leveling phase, an average of 8 months
  Incisal mandibular plane angle

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Forero, Principal Investigator

IPD SHARING:
Plan to Share IPD: No